CLINICAL TRIAL: NCT05719077
Title: Study 3. Pilot Testing Feasibility, Acceptability, and Preliminary Efficacy of a Dementia-Enhanced Training and Tool for Home Hospice Clinicians in a Clinical Setting.
Brief Title: Pilot Testing Dementia-Enhanced Training and Tool for Home Hospice Clinicians
Acronym: EDITH-HC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elizabeth A. Luth, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2021001817; R00AG065624 (NIH)
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease and Related Dementias
Keywords: Dementia; End of life; Hospice; Caregiver Burden; Caregiving
MeSH Terms: conditions — Alzheimer Disease; Dementia; Death; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Nurses and social workers are organized into interdisciplinary teams (IDTs) based on geographic location. Patients and families in those geographic are assigned to clinicians' individual caseloads. The investigators will randomize up to 14 IDTs of 6-8 clinicians each to the intervention and control groups. Six teams will be randomized at the beginning of the study. The remaining 8 teams will be adaptively randomized as they enter the study to maintain balance between the number of Black and White family caregiver participants in each arm. Family caregivers will be assigned to the same group (intervention or control) as the clinician they are assigned to. IDT assignment to intervention and control groups will be balanced based on characteristics including patients' racial/ethnic group membership and neighborhood socioeconomic status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Clinicians in intervention group will watch a series educational and instructional videos and use caregiver burden assessment tool up to four times during regular home visits with family caregivers of home hospice patients living with dementia. Clinicians will be assessed for changes in knowledge regarding dementia caregiving (secondary outcome). Family caregivers will be assessed for changes in caregiver burden (primary outcome) and preparedness and self-efficacy (exploratory outcomes).
  Interventions: Behavioral: EDITH-HC
- Control Group (Other): Clinicians in control group will listen to a presentation on outcomes for home hospice patients living with dementia. Clinicians will be assessed for changes in knowledge regarding dementia caregiving (secondary outcome). Family caregivers will be assessed for changes in caregiver burden (primary outcome) and preparedness and self-efficacy (exploratory outcomes).
  Interventions: Behavioral: EDITH-HC

INTERVENTIONS:
Behavioral: EDITH-HC — This study tests feasibility and acceptability of implementing a tool and training in a clinical practice and the preliminary efficacy of training materials to enhance hospice clinicians' knowledge of dementia-related caregiving issues at end of life and a tool for clinicians to use to address caregiving issues related to dementia at end of life.

SUMMARY:
The purpose of this study is to pilot test the feasibility, acceptability, and preliminary efficacy of a clinically useful, inclusive dementia-enhanced training and tool for use by home hospice clinicians to improve care and support for Black and White patients with dementia and their family caregivers. The investigators expect family caregivers of clinicians in the intervention group will report less caregiver burden (primary outcome) than caregivers of clinicians in the control group. The investigators expect that, compared to clinicians in the control group (usual care), clinicians in the intervention group (receive the training and use the tool) will demonstrate more knowledge of dementia-related caregiving issues (secondary outcomes). In exploratory analyses, the investigators expect family caregivers will report greater self-efficacy and preparedness, and that patients of clinicians in the intervention group will experience fewer live discharges than family caregivers of patients of clinicians in the control group.

DETAILED DESCRIPTION:
For this aim, the investigators will conduct a randomized pilot study to determine the feasibility and acceptability of implementing the training and tool in clinical practice compared to usual care with 40 clinicians (20 intervention, 20 control) and 160 Black and white FCG (80 intervention, 80 control). The investigators will also determine preliminary efficacy of the training and tool. Outcomes include feasibility and acceptability of the intervention, reducing FCG burden (primary outcome), improving clinician knowledge and confidence (secondary outcomes) and increasing FCG preparedness and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals are not excluded from this study based on gender.
* Based on proportion of hospice workforce and family caregivers that are female, we expect 70%-80% of participants will be female.
* Nurse, social worker, or family member who provides care to persons(s) living with dementia enrolled in home hospice care.
* 19-90 years old.
* Can complete data collection in English.
* Family Caregivers: identify as White or Black/African American.

Exclusion Criteria:

* Participant is less than 19 years old or older than 90 years old.
* Does not provide care to person(s) living with dementia enrolled in home hospice.
* Cannot complete data collection in English.
* Family Caregiver does not identify as White or Black/African American.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
Family Caregiver Burden | Baseline and through first subsequent hospice visit, an average of 8 weeks
  The investigators will assess this outcome using the validated, 12-item Zarit Caregiver Burden Inventory. The investigators will assess changes in reported caregiver burden between baseline and the frist subsequent hospice visit and compare differences in changes between the intervention and control groups. Because family caregiver participants are relatives of hospice patients that may die (at which point they will no longer be receiving home visits from nurses and social workers), the investigators expect that many participants will not complete all four time points of data collection.

SECONDARY OUTCOMES:
Clinician knowledge of dementia-related issues at end of life | Baseline and through training completion, an average of 4 weeks
  The investigators will assess clinician knowledge of dementia-related issues at end of life using a revised Dementia Knowledge Assessment Scale and assessment questions that are tailored to the content of the training. The investigators will assess changes in reported knowledge between baseline and after completing the training. The investigators will compare differences in changes between clinicians receiving the training (intervention) and those receiving a presentation on patterns of hospice outcomes for persons living with dementia (control).

OTHER OUTCOMES:
Family caregiver self-efficacy (exploratory) | Baseline and through first subsequent hospice visit, an average of 8 weeks
  The investigators will assess caregiver self-efficacy using the validated, 8-item Caregiver Self-Efficacy Scale (CSES). The investigators will assess changes in caregiver self-efficacy between baseline and the first subsequent hospice visit and compare differences in changes between the intervention and control groups. The same issues due to attrition described in 1. Family Caregiver burden above also apply here.
Family caregiver preparedness (exploratory) | Baseline and through first subsequent hospice visit, an average of 8 weeks
  The investigators will assess caregiver preparedness for dementia caregiving using a single-item question about the extent to which caregivers feel prepared to provide care to their loved one and the 9-item Preparedness Scale of the Family Care Inventory. The investigators will assess changes at baseline and the first subsequent hospice visit and compare differences in changes between the intervention and control groups. The same issues due to attrition described in 1. Family Caregiver burden above also apply here.
Patient hospice discharge status (exploratory) | 3 months post-intervention, 6 months post-intervention
  The investigators will assess patient status upon hospice discharge as either deceased or alive. The investigators will assess patient discharge status as reported in the electronic hospice records. The investigators will compare discharge status of hospice patients with study-enrolled caregivers between intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Luth, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers Univeristy, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No